CLINICAL TRIAL: NCT03558100
Title: A Nonrandomized Controlled Trial of an Obstacle Crossing Intervention for Adults Before Bariatric Surgery
Brief Title: Reducing Fall Risks for Adults With Obesity
Acronym: ObesityFalls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Simone V. Gill, Associate Professor, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3820E; R03AR066344-01A1 (NIH)
Record Dates: First submitted 2018-05-25; First posted 2018-06-15 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Bariatric Surgery Candidate; Gait, Unsteady
Keywords: obesity; gait; bariatric surgery; walking; obstacles
MeSH Terms: conditions — Obesity; Gait Disorders, Neurologic | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reducing Fall Risks in Obesity (Experimental): Adults with obesity will be asked to perform the obstacle crossing intervention for adults with obesity for reducing falls risk. This will involve crossing obstacles of different heights under five conditions: initial baseline walking on flat ground, crossing three obstacle heights, and final baseline walking on flat ground for a total of 25 trials. Spatio-temporal gait parameters will be collected using a gait carpet and body-worn sensors.
  Interventions: Behavioral: Obstacle crossing intervention for adults with obesity

INTERVENTIONS:
Behavioral: Obstacle crossing intervention for adults with obesity — The obstacle crossing intervention will be done for reducing falls risks in obesity. The intervention will provide gait practice to individuals with obesity who are eligible for and prior to weight loss surgery.

SUMMARY:
The objective of the clinical study was to examine if practice could improve walking patterns associated with fall risks before patients with obesity underwent weight loss surgery. We hypothesized that patients would show improvements in their walking after completing the intervention. For the intervention, patients walked under five conditions: on flat ground at the beginning of the study, crossing three obstacle heights, and on flat ground at the end of the study for a total of 25 times.

DETAILED DESCRIPTION:
Obesity has a negative impact on aspects of walking associated with fall risks. After weight loss surgery, adults show improvements in walking. However, those who undergo surgery still show deficits in walking and an additional group of individuals do not undergo the procedure. Our objective was to examine if practice could improve gait patterns associated with fall risks before patients underwent weight loss surgery. Adults with obese body mass index between 30 to 60 years old who were eligible to undergo the Roux-en-Y weight loss surgery procedure walked under five conditions: initial baseline walking on flat ground, crossing three obstacle heights, and final baseline walking on flat ground for a total of 25 trials. Spatio-temporal gait parameters were collected using a gait carpet and body-worn sensors. The GAITRite mat was a 4.9 m long x 0.6 m wide pressure-sensitive mat with a temporal resolution of 120 Hz and a spatial resolution of 1.3 cm. LEGSysTM includes five wearable sensors containing triaxial gyroscopes, accelerometers, and magnetometers. Dependent variables selected included velocity (cm/s), cadence (steps/minute), step length (distance between consecutive steps), step width (lateral distance between feet), single limb support time (amount of time spent on one leg during the walking cycle), and double limb support time (amount of time spend on two legs during the walking cycle).

ELIGIBILITY:
Inclusion Criteria:

* between 30 and 60 years old
* eligible to undergo Roux-en-Y gastric bypass surgery
* walk independently without assistive devices

Exclusion Criteria:

* scheduled to undergo knee surgery
* receiving dialysis
* being treated for cancer

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Velocity (cm/s) | The change from baseline velocity (cm/s) at 12 months
  walking speed

SECONDARY OUTCOMES:
Cadence (steps per minute) | The change from baseline cadence (steps per minute) at 12 months
  steps per minute
Step width (cm) | The change from baseline step width (cm) at 12 months
  lateral distance between feet
single limb support time (msec) | The change from baseline single limb support time (msec) at 12 months
  time spent balancing on one leg
double limb support time (msec) | The change from baseline double limb support time (msec) at 12 months
  time spent balancing on both legs
step length (cm) | The change from baseline step length (cm) at 12 months
  distance between consecutive steps

CONTACTS AND LOCATIONS:
Overall Officials: Simone V Gill, Principal Investigator — Boston University Charles River Campus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gill SV, Walsh MK, Pratt JA, Toosizadeh N, Najafi B, Travison TG. Changes in spatiotemporal gait patterns during flat ground walking and obstacle crossing 1 year after bariatric surgery. Surg Obes Relat Dis. 2016 Jun;12(5):1080-1085. doi: 10.1016/j.soard.2016.03.029. Epub 2016 Mar 30. PMID 27320220